CLINICAL TRIAL: NCT06189911
Title: The Risk Factors for Perioperative Blood Transfusion in Open Liver Resection, a Retrospective Cohort Study Development of a Transfusion Scoring System to Predict the Requirement for Perioperative Blood Transfusion in Open Liver Resection
Brief Title: Perioperative Blood Transfusion in Open Liver Resection
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Warangkana Lapisatepun, Assistant professor, Chiang Mai University
Other Study IDs: ANE-2564-08020
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Blood Loss, Postoperative
Keywords: liver resection; risk factors; blood transfusion; scoring system
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transfused: Group of patients who received perioperative blood transfusions which was defined as the transfusion of packed red cells during the operation and 48 hours after surgery.
  Interventions: Procedure: Open liver resection
- non-transfused: Group of patients who did not received perioperative blood transfusions
  Interventions: Procedure: Open liver resection

INTERVENTIONS:
Procedure: Open liver resection — The definitions of liver resection and the type of hepatectomy were aligned with the anatomic classification of the Brisbane 2000 Terminology

SUMMARY:
This observational study is specifically designed to identify the pre-operative risk factors that significantly contribute to perioperative packed red cell transfusions in open liver resection procedures.

The main question it aims to answer are:

1. What are the risk factors of peri-operative blood transfusion in open liver resection procedures
2. What are the difference outcomes between patients who receive blood transfusion and the other group.

Researcher will compare perioperative factor and post operative outcomes between transfused and non-transfused group

DETAILED DESCRIPTION:
After approval of the study protocol from the institutional review board of Chiangmai University (Approval number: ANE-2564-08020), we performed a retrospective review of all patients who underwent an elective open liver resection in our specialized hepato-biliary center from January 2006 through December 2017. This retrospective inquiry comprised 808 patients.

The data was systematically retrieved from electronic medical records. Baseline characteristics including age, gender, body mass index (BMI), co-morbidity, American Society of Anesthesiologists (ASA) classification, diagnosis, hepatitis profile, Child-Pugh classification, cirrhosis, the largest tumor size, previous liver resection, and pre-operative laboratory investigations were collected.

The following intra-operative data were collected: type of liver resection, hilar resection, vascular reconstruction, volume and type of fluid administration, estimated blood loss, packed red cell and blood product transfusion, and operation time. The definitions of liver resection and the type of hepatectomy were aligned with the anatomic classification of the Brisbane 2000 Terminology

ELIGIBILITY:
Inclusion Criteria:

* All genders age above 18 year old who underwent open liver resection from 2006-2017
* Elective open liver resection

Exclusion Criteria:

* Patients who death during the course of a surgical operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who underwent an elective open liver resection in our specialized hepato-biliary center from January 2006 through December 2017
Sampling Method: Non-Probability Sample
Enrollment: 1201 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
the pre-operative risk factors of perioperative packed red cell transfusions in open liver resection procedures. | the transfusion of packed red cells during the operation and 48 hours after surgery
  Significant risk factors for perioperative blood transfusion were determined by factors with a p-value < 0.05 derived from the multivariable logistic regression analysis. This analysis facilitated adjustments for potential confounders to identify the independent risk factors associated with perioperative blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Warangkana Lapisatepun, M.D., Principal Investigator — Chiang Mai University

IPD SHARING:
Plan to Share IPD: No
Did not state about IPD sharing in the proposal which proposed to institutional review board.